CLINICAL TRIAL: NCT03157752
Title: Evaluation of the Satisfaction of Patients With Conization Under Local Anesthesia, Prospective Study
Brief Title: Evaluation of the Satisfaction of Patients With Conization Under Local Anesthesia
Acronym: ESCAL
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Collaborators: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL17_0145
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-05

CONDITIONS: Local Anaesthetic Complication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Quality of life questionnaire — Quality of life questionnaire

SUMMARY:
In France, screening involves a routine test of papanicolaou in women aged 25 to 65 years. In the case of an abnormal Pap smear discovery, the diagnostic strategy is based in most cases in colscopy to allow cervical biopsies if necessary to obtain a histological diagnosis of high quality cervical intraepithelial neoplasia (CIN) (2- 3) which, if persistent, can cause cervical cancer. Their results, also in the case of the persistence of a low-level lesion or of a cyto-histological discordance, indicate conization. Conization is a procedure performed by resection of the diathermic grip, allowing a simple and fast gesture compatible with a load under local anesthesia. In order to simplify the overall cost of the patient, more and more conizations of Montpellier and Nimes take place under local anesthesia. .

The main objective of our study is to evaluate the overall satisfaction of patients in the case of conisation under local anesthesia.

The goal is to promote local anesthesia for the management of congested patients, which simplifies overall management, reduces cost and reduces complications associated with general anesthesia.

DETAILED DESCRIPTION:
In France the screening is on the regular realization of a papanicolaou test (Pap smear or Pap test) in women aged 25 to 65 years. In the event of abnormal Pap smear discovery, the diagnostic strategy is based in most cases on colscopy to allow for cervical biopsies if necessary to obtain a histological diagnosis for cervical intraepithelial neoplasia (CIN ) High grade (2-3) which, if persistent, may cause cervical cancer. Their findings, also in the case of persistence of low-grade lesion or cyto-histological discordance, indicate conization. The conization is an intervention realized by resection to the diathermic handle, allowing a simple and fast gesture compatible with a charge under local anesthesia. With a view to simplify the overall cost of the patient, more and more conizations of the Montpellier and Nimes are carried out under local anesthesia. A retrospective study found a good overall satisfaction of the patients with conisation under local anesthesia, it is interesting to continue this study by an evaluation of the patient's satisfaction in the prospective way, including validated rankings and to allow a risk assessment And the persistence of lesions.

The main objective of our study is to evaluate the overall satisfaction of the patients in the case of conducting conization under local anesthesia. Secondary endpoints are preoperative anxiety assessed using the Visual Analog Scale (EVA) And the Amsterdam Preoperative Anxiety and Information Scale (APAIS) score, the occurrence of complications during the procedure, surgeon satisfaction, anesthesia tolerance using the Iowa Satisfaction with Anesthesia Scale score (ISAIS), and finally A follow-up at 3 months evaluation of secondary complications, margins of resections and persistence of lesions.

This is a prospective multi-centric study (CHU Nîmes and Montpellier). During the day hospitalization, a questionnaire of satisfaction will be given to the patient. The primary outcome measure is the overall satisfaction of the patient assessed as a question. Secondary endpoints are preoperative anxiety assessed using the visual analog scale (EVA) and the Amsterdam Preoperative Anxiety and Information scale (APAIS) score, the occurrence of complications during gesture, satisfaction of the surgeon , Tolerance of anesthesia using the ISAS score, and finally a 3-month follow-up to evaluate secondary complications, resection margins and lesions persistence. Currently the only study on the subject is a retrospective study of 70 subjects. This study reported a proportion of patients with little or no satisfaction of 11.4%. Recruiting 80 patients will confirm this rate with an accuracy of +/- 7%.

The questionnaire will be given on the day of surgery and completed before surgery, immediately after surgery and before final discharge. Secondarily, the data will be supplemented during a postoperative control visit at 3 months of the intervention. The expected duration of the inclusions is 10 months with follow-up at 3 months

The aim is to promote local anesthesia for the management of congested patients, thus simplifying the overall management, reducing the cost and reducing the complications associated with general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* Patient requiring conization on the CHU of Montpellier or Nîmes and having chosen a local anesthesia.
* Informed and not opposed to participate in this research

Exclusion Criteria:

* Contra-indication to local anesthesia

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Patient requiring conization on the CHU of Montpellier or Nîmes and having chosen a local anesthesia.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2017-05-31 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Patient satisfactio | 1 day
  Overall satisfaction of the patient, evaluated by the completion of a questionnaire on the day of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Elsa MARIS, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC